CLINICAL TRIAL: NCT03695731
Title: Influence of Diabetic Neuropathy on Activation of Brown Adipose Tissue
Acronym: DIA-BAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Doctor Giacomo Gastaldi (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Sponsor-Investigator, Doctor Giacomo Gastaldi, Principal investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14-170 (PB_2018-00258)
Record Dates: First submitted 2018-09-26; First posted 2018-10-04 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: diabetes; brown adipose tissue; energy expenditure; glycemic control; neuropathy; 18F-FDG PET-RMI
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients without Neuropathy (Experimental): activation of cold induced brown adipose tissue
  Interventions: Procedure: cold induced activation of brown adipose tissue
- Patients with Neuropathy (Experimental): activation of cold induced brown adipose tissue
  Interventions: Procedure: cold induced activation of brown adipose tissue

INTERVENTIONS:
Procedure: cold induced activation of brown adipose tissue — cold exposure wearing a cold life jacket

SUMMARY:
Influence of diabetic neuropathy on cold induced brown adipose tissue in type 1 diabetic patients.

DETAILED DESCRIPTION:
The prevalence of type 1 diabetes has been steadily increasing for about 20 years. Despite therapeutic progress, between 20 and 65% of people with diabetes develop diabetic neuropathy, resulting in increased morbidity and mortality.

Diabetic neuropathy is not limited to sensitive pain in the lower limbs. It also affects the fibres of the autonomic nervous system (ANS), which results in systemic complications, often disabling (erectile dysfunction, dysidrosis, gastroparesis, orthostatism, etc.) and a probable alteration in the body's thermogenic capacities, although this possibility has not been studied in humans. In rodents, it is possible to activate induced thermogenesis via central stimulation of the ANS or to inactivate it, which promotes the development of obesity and greater insulin resistance. This knowledge is based on cellular and animal models that have identified the bio-molecular mechanisms that give brown adipose tissue (BAT) the ability to dissipate energy in the form of heat.

Induced thermogenesis is mediated by decoupling proteins 1 (DCS-1) located on the mitochondrial inner membrane of the TAB. DCS-1 decouple oxidative phosphorylation from ATP production, dissipating the proton gradient. The activation of UCP1 is particularly influenced by the sympathetic system and more particularly by catecholamines which will bind to ß3 adrenergic receptors (Rß3). In humans, the persistence of active areas of TAB has recently been demonstrated by positron emission tomography (PET) imaging using a glucose analogue radiotracer, 18F-Fluoro-Deoxy-Glucose (18F-FDG), coupled with the scanner (CT). Recently, it has been shown that the use of 18F-FDG PET coupled with magnetic resonance (MRI) is equally effective in differentiating TAB from white fat tissue with less patient irradiation. The activity of the TAB is estimated using the measurement of SUV (standard uptake value) which represents the total glycolytic activity of the tissue and is also commonly referred to as the total metabolic volume. It has been shown in humans that TAB activity is inversely correlated with body mass index and age and positively correlated with exposure to cold and stress levels[6]. Among diabetics, the data are disparate but the spontaneous prevalence of TAB appears to be reduced compared to the general population (1.1% vs 7.5%). To date, no studies have investigated a possible link between the decrease in TAB activity observed in diabetics and the presence of autonomic neuropathy, which is a common and often under-diagnosed complication of diabetes.

The main purpose of this study is to evaluate whether the activity and distribution of TAB in patients with diabetes is influenced by the presence of diabetic neuropathy. On the other hand, if the existence of diabetic neuropathy influences energy expenditure in the event of exposure to cold. Finally, whether any differences in the activity and distribution of TAB could be related to changes in the central nervous system.

The investigators plan to include a total of 24 patients with type 1 diabetes and separate them into 2 groups: group A; no neuropathic complications and group B; presence of neuropathy. All patients will be characterized in terms of clinical, metabolic and energy expenditure. The activity of the TAB will be evaluated through the use of 18F-FDG PET/IRM imaging, after a cold stimulation protocol (refrigerated jacket) in order to activate the TAB in a homogeneous manner among the participants.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 diabetes
2. Patients who can understand the issue of this study and who are able to decide for themselves whether or not to participate in the study.
3. Adult patient (>18 years old)
4. Informed Consent form signed
5. Differentiated inclusion:

   * Group A: absence of neuropathy
   * Group B: significant neuropathy

Exclusion Criteria:

1. Treatment with beta-blockers
2. Alcohol consumption(> 50 gr/week)
3. Allergy to 18F-FDG
4. Participation in another clinical study (4 weeks prior to entry) that may influence the activity of brown adipose tissue
5. Pregnancy
6. Exposure to ionizing radiation greater than or equal to 5 mSv during the year preceding the PET-RMI planned in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-10-15 (Estimated); Study Completion 2019-10-15 (Estimated)

PRIMARY OUTCOMES:
brown adipose tissue activation | 120 minutes after cold exposure
  PET- MRI measurement (SUVR)

SECONDARY OUTCOMES:
Energy expenditure | before and 120 minutes after cold exposure
  indirect calorimetry measurement

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Gastaldi, Dr., Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided